CLINICAL TRIAL: NCT04893941
Title: A Randomized, Double Blind, Placebo-controlled, Multiple Dose Escalation, Phase Ib/IIa Study to Evaluate the Safety, Tolerance, PK, PD, Immunogenicity and Preliminary Efficacy of Subcutaneously CM310 in Moderate-severe AD Subjects.
Brief Title: Dose Escalation Trial of CM310 in Patients With Moderate-to-Severe Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310AD001
Record Dates: First submitted 2021-04-25; First posted 2021-05-20 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CM310 75mg arm (Experimental): 75mg for 3 doses, every 2 weeks, SC
  Interventions: Drug: CM310
- CM310 150mg arm (Experimental): 150mg for 3 doses, every 2 weeks, SC
  Interventions: Drug: CM310
- CM310 300mg arm (Experimental): 300mg for 3 doses, every 2 weeks, SC
  Interventions: Drug: CM310
- CM310 600(1st)+300mg(2nd,3rd) arm (Experimental): 600mg for 1st dose, and then 300 mg for 2nd and 3rd doses, every 2 weeks, SC
  Interventions: Drug: CM310
- placebo arm (Placebo Comparator): placebo for 3 doses, every 2 weeks, SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM310 — IL-4Rα monoclonal antibody
  Arms: CM310 150mg arm; CM310 300mg arm; CM310 600(1st)+300mg(2nd,3rd) arm; CM310 75mg arm
Drug: Placebo — Placebo
  Arms: placebo arm

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled multiple dose escalation study to evaluate the safety, tolerance, PK, PD, immunogenicity and preliminary efficacy of subcutaneously CM310 in moderate-severe AD subjects.

DETAILED DESCRIPTION:
The study consists of 3 periods, a up-to-4-week Screening Period, a 4-week randomized Treatment Period and a 8-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as AD for at least 12 months before Screening, with below requirements: 1)EASI score ≥16 at Screening and Baseline; 2) IGA score ≥3 (0-5 points scale) at Screening and Baseline; 3) ≥10% BSA of AD involvement at Screening and Baseline; 4) Pruritus NRS average score ≥3 at Baseline.
* Inadequate response to topical medications.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Concurrent disease/status which may potentially affect the efficacy/safety judgement.
* Organ dysfunction.
* Pregnancy.
* Other.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Safety parameters (e.g., Incidence of AE, abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing) | Baseline to Week 12
  Incidence of AE, abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Peak concentration (Cmax) | Baseline to Week 12
  Peak concentration (Cmax)
Pharmacokinetics parameter: Area under the plasma concentration-time curve from 0 to ∞ (AUC0-∞) | Baseline to Week 12
  Area under the plasma concentration-time curve from 0 to ∞ (AUC0-∞)
Pharmacokinetics parameter: Area under the plasma concentration-time curve from 0 to t (AUC0-t) | Baseline to Week 12
  Area under the plasma concentration-time curve from 0 to t (AUC0-t)
Pharmacokinetics parameter: Clearance rate (CL/F) | Baseline to Week 12
  Clearance rate (CL/F)
Pharmacodynamics parameters: Serum Thymus and activation regulated chemokine (TARC) | Baseline to Week 12
  Serum Thymus and activation regulated chemokine (TARC), total IgE level and blood eosinophil count (EOS)
Pharmacodynamics parameters: Blood eosinophil count (EOS) | Baseline to Week 12
  Blood eosinophil count (EOS)
Pharmacodynamics parameters: Total IgE level | Baseline to Week 12
  Total IgE level
Immunogenicity: Proportion of subjects with anti-drug antibody (ADA) | Baseline to Week 12
  Proportion of Participants with anti-drug antibody (ADA)
Preliminary efficacy: Proportion of subjects with IGA 0 or 1 | Baseline to Week 12
  Proportion of subjects with Investigator's Global Assessment (IGA, on a 6-point scale, range from 0-5 point, higher scores mean a worse disease severity) 0 or 1
Preliminary efficacy: Proportion of subjects with a reduction of IGA from baseline of ≥ 2 points | Baseline to Week 12
  Proportion of subjects with a reduction of IGA from baseline of ≥ 2 points
Preliminary efficacy: Proportion of subjects with IGA 0 or 1 and a reduction of IGA from baseline of ≥ 2 points | Baseline to Week 12
  Proportion of subjects with IGA 0 or 1 and a reduction of IGA from baseline of ≥ 2 points
Preliminary efficacy: Proportion of subjects with EASI-50 | Baseline to Week 12
  Proportion of subjects with The Eczema Area and Severity Index(EASI)-50 (≥50 percent improvement from baseline)
Preliminary efficacy: Proportion of subjects with EASI-75 | Baseline to Week 12
  Proportion of subjects with EASI-75 (≥75 percent improvement from baseline)
Preliminary efficacy: Proportion of subjects with improvement (reduction) of pruritus NRS from baseline | Baseline to Week 12
  Proportion of subjects with improvement (reduction) of pruritus Numerical Rating Scale(NRS) from baseline; The range of NRS is from 0 (no itch)-10 (worst imaginable itch)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Second Hospital, Wuxi, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Shanghai Skin Disease Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Zhang W, Xu Y, Dong L, Sun Y, Jia Y, Li Z, Chen B, Hou J, Zhang J. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Stapokibart in Healthy Volunteers and Adult Subjects with Atopic Dermatitis. Adv Ther. 2024 Jul;41(7):2953-2965. doi: 10.1007/s12325-024-02887-w. Epub 2024 Jun 4. PMID 38833140